CLINICAL TRIAL: NCT05046613
Title: A Prospective, Registry-based, Observational Study to Assess Maternal, Fetal and Infant Outcomes Following Exposure to Rimegepant: The Migraine Observational Nurtec Pregnancy Registry (MONITOR)
Brief Title: Observational Study to Assess Maternal, Fetal and Infant Outcomes Following Exposure to Rimegepant
Acronym: MONITOR
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: PPD, Part of Thermo Fisher Scientific (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV3000-402; C4951005 (Other: Alias Study Number)
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine, Migraine Headache, Pregnant, Pregnancy, Infant
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with migraine exposed to Rimegepant: Pregnant women with a diagnosis of migraine who are exposed to rimegepant at any time during pregnancy or just prior to pregnancy (up to 3 days prior to conception)
  Interventions: Other: Rimegepant
- Pregnant women with migraine not exposed to Rimegepant: Pregnant women with a diagnosis of migraine who are not exposed to rimegepant (up to 5 product half-lives prior to conception) but who may be exposed to other products for the treatment/prevention of migraine at any time during pregnancy or just prior to pregnancy
  Interventions: Other: Not taking Rimegepant

INTERVENTIONS:
Other: Rimegepant — 75mg
  Groups: Pregnant women with migraine exposed to Rimegepant
Other: Not taking Rimegepant — No rimegepant
  Groups: Pregnant women with migraine not exposed to Rimegepant

SUMMARY:
The purpose of the study is to evaluate fetal, maternal, and infant outcomes through 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with migraine exposed to rimegepant: a diagnosis of migraine and at least 1 dose of rimegepant during pregnancy or just prior to pregnancy (up to 3 days prior to conception)
* Pregnant women with migraine unexposed to rimegepant: a diagnosis of migraine and no exposure to Rimegepant before or during pregnancy

Exclusion Criteria:

• Women exposed to other calcitonin gene-related peptide (CGRP)antagonists (e.g., ubrogepant), CGRP monoclonal antibodies, or ditans (e.g., lasmiditan) at any time during pregnancy or just prior to pregnancy

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include pregnant women of any age within the US with migraine who were treated with rimegepant as part of routine care at any time during pregnancy or just prior to pregnancy (up to 3 days prior to conception), as well as pregnant women with migraine not exposed to rimegepant before or during pregnancy.
Sampling Method: Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2034-04-30 (Estimated); Study Completion 2034-04-30 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformation (birth defect) | Annually beginning April 2022
  Healthcare provider report through the registry

SECONDARY OUTCOMES:
Minor congenital malformation | Annually beginning April 2022
  Healthcare provider report through the registry
Gestational hypertension | Annually beginning April 2022
  Healthcare provider report through the registry
Pre-eclampsia | Annually beginning April 2022
  Healthcare provider report through the registry
Eclampsia | Annually beginning April 2022
  Healthcare provider report through the registry
Gestational diabetes | Annually beginning April 2022
  Healthcare provider report through the registry
Spontaneous abortion | Annually beginning April 2022
  Healthcare provider report through the registry
Stillbirth | Annually beginning April 2022
  Healthcare provider report through the registry
Elective termination | Annually beginning April 2022
  Healthcare provider report through the registry
Preterm birth | Annually beginning April 2022
  Healthcare provider report through the registry
Small for gestational age | Annually beginning April 2022
  Healthcare provider report through the registry
Postnatal growth deficiency | Annually beginning April 2022
  Healthcare provider report through the registry
Infant developmental delay | Annually beginning April 2022
  Healthcare provider report through the registry

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Evidera, a PPD business unit, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-402
- See also: Nurtec Pregnancy Registry — https://nurtecpregnancyregistry.com/